CLINICAL TRIAL: NCT06256523
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ib/IIa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of GZR18 Injection in Chinese Adult Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: A Study of GZR18 Injection in Chinese Adult Patients With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GLP-CH2001
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR18 (Experimental): GZR18 injection s.c.
  Interventions: Drug: GZR18
- Placebo (Placebo Comparator): Placebo injection s.c.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GZR18 — 0.5mg-13mg
  Arms: GZR18
Other: Placebo — administered the same volume as GZR18
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase Ib/IIa clinical study in Chinese patients with type 2 diabetes mellitus (T2DM) inadequately controlled with diet and exercise and/or treated with irregular use of antidiabetic drugs to evaluate the safety, tolerability, pharmacokinetics and efficacy of GZR18 injection in adult subjects with T2DM. This study is divided into Part A and Part B, which are to be conducted simultaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults, male and female, aged 18-65 years (both inclusive; subject to the date of signing of ICF).
2. Diagnosis of type 2 diabetes mellitus according to the diagnostic and classification criteria for diabetes mellitus issued by the World Health Organization (WHO) in 1999.
3. Patients with type 2 diabetes mellitus (T2DM) inadequately controlled with diet and exercise and/or treated with irregular use of antidiabetic drugs.
4. Hemoglobin A1c (HbA1c) ≥ 7.0% and ≤ 10 % at screening;
5. Body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 35 kg/m2 at screening.
6. Those who have no birth and sperm donation plans, and voluntarily take effective contraceptive measures from the signing of ICF to 3 months after the last dose. A negative pregnancy test for women of childbearing potential at screening.
7. Fully understanding the study objectives, the nature of the study, methods used and adverse reactions that may occur in the study, willing to enter the study and sign the ICF, and capable of communicating well with the investigator, and understanding and abiding by the requirements of the study.

Exclusion Criteria:

1. Diabetes mellitus other than T2DM, such as type 1 diabetes mellitus.
2. Fasting C-peptide < 0.3 nmol/L.
3. Use of any DPP-4 inhibitors, insulin secretagogues such as sulfonylureas, TZDs and/or GLP-1 analogs within 3 months prior to screening.
4. Continuous insulin use for more than 14 days within 1 year prior to screening (time of insulin use for gestational diabetes mellitus is excluded from this limit).
5. Treatment with growth hormone, diuretics, etc., that may affect insulin levels as judged by the investigator within 6 months prior to screening.
6. Immunoserologic panel test results [infection screening tests for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), and Treponema pallidum antibody] assessed by the investigator as abnormal and clinically significant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events | 29 weeks
Changes from baseline in hemoglobin A1c (HbA1c) at the end of the study | 26 weeks

SECONDARY OUTCOMES:
Trough concentrations of GZR18 following consecutive doses | 26 weeks
HbA1c control rate (proportions of subjects with HbA1c < 6.5 % and HbA1c < 7.0 %) | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhao, Ph.D, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, China